CLINICAL TRIAL: NCT01277003
Title: To Investigate the Therapeutic Effect of Aculife Magnetic Therapist on Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: China Medical University Hospital, China Medical University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0994266G
Record Dates: First submitted 2011-01-13; First posted 2011-01-14 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2010-11

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aculife Magnetic Wave Therapist (Experimental): patients with carpal tunnel syndrome treated with Aculife
  Interventions: Device: Aculife Magnetic Wave Therapist
- TENS (Active Comparator): patients with carpal tunnel syndrome treated by TENS
  Interventions: Device: TENS

INTERVENTIONS:
Device: Aculife Magnetic Wave Therapist — two therapeutic points, each for 15 minutes
  Arms: Aculife Magnetic Wave Therapist
Device: TENS — tow therapeutic points, each for 15 minutes
  Arms: TENS

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common compressive focal mononeuropathy seen in clinical practice. Patients commonly experience a constellation of symptom complex brought on by compression of the median nerve as it traverse through the carpal tunnel. When compression of the nerve occurs, ischemia and mechanical disruption of nerve function may result. Pathological analysis shows a constellation of nerve injuries. Until now, no satisfactory conservative treatment method. Local steroid injections or oral steroids may result in initial relief, but relapses are frequent and have much side effects, which preclude their routine use for CTS. Full time wrist splints are claimed effective, but compromise hand function and daily activities. There are reasonable studies showing relief of pain with acupuncture on diverse pain conditions. However the therapeutic efficacy of acupuncture in CTS was less convincing in the past. Until recent decade, some case reports and few prospective studies reported the therapeutic effect of acupuncture in CTS. Other study also reported that low-level laser and microamperes transcutaneous electrical nerve stimulation (TENS) are effective in improvement of clinical outcome of patients with CTS. Another report suggested that TENS should be considered for the treatment of painful diabetic peripheral neuropathy. Therefore, the investigators perform this study to evaluate the effect of Aculife Magnetic Wave Therapist (a battery operated device with a probe electrode which contains magnetic elements that transform the oscillating current into an electromagnetic wave to stimulate the acupuncture points, simulate the effect of electroacupuncture ) on CTS and compared with that of Transcutaneous Electrical Nerve Stimulation(TENS). After at least 4 weeks treatment ( at least 16 treatment sessions) the therapeutic effects will be evaluated by comparison of symptom severity score, electrophysiological study, sonographic morphology study or magnetic resonance imaging study, before and after treatment, and between the different groups.

ELIGIBILITY:
Inclusion Criteria:

* electrodiagnostic study confirmed with carpal tunnel syndrome
* clinical symptom related to carpal tunnel syndrome

Exclusion Criteria:

* hypothyroidism, gout, systemic lupus erythematosus, rheumatoid arthritis, diabetes mellitus, chronic renal failure, acromegaly, polyneuropathy, brachial plexopathy, proximal median nerve entrapment, deficiency neuropathy (vitamine 2, B12, ect.), drug usage that may cause neuropathy, any surgery for peripheral nerve in the upper limb such as carpal tunnel surgical release, history of trauma in the upper limb such as wrist fracture, or having pregnancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
nerve conduction study | after at least four weeks treatment (at least 16 treatment sesstions)

SECONDARY OUTCOMES:
questionnaire | after at least four weeks treatment ( at least 16 treatment sesstions)

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Taichung, Taiwan, Taiwan